CLINICAL TRIAL: NCT02821520
Title: Efficacy and Safety of Initial Versus Delayed Verteporfin Photodynamic Therapy in Combination With Conbercept in Patients With Symptomatic Polypoidal Choroidal Vasculopathy
Brief Title: Initial Versus Delayed PDT Combination With Conbercept in PCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiaoling Liu, professor, The Eye Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y-2016020
Record Dates: First submitted 2016-06-25; First posted 2016-07-01 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal Choroidal Vasculopathy; Photodynamic Therapy; Conbercept; Efficacy; Safety; vascular endothelial growth factor
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — KH902 fusion protein; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial PDT combination with Conbercept (Experimental): 1. Conbercept 0.5 mg(0.05ml): Administered at baseline, and then PRN based on retreatment criteria monthly from month 1 to 11.
  2. PDT: PDT with verteporfin is administered at baseline and then PRN PDT combination with conbercept injection based on retreatment criteria from month 3 to 11.
  PDT treatment must be administered within 7 days after the injection. If same day treatment of conbercept and PDT is performed, conbercept injection is to be administered at least 2 hours after the PDT.
  PDT should cover the whole area of polyps and branch vascular net (BVN).The PRN PDT retreatment intervals should be no less than 3 months.
  Interventions: Drug: conbercept; Procedure: Initial PDT
- Delayed PDT combination with Conbercept (Active Comparator): 1. Conbercept 0.5 mg(0.05ml): Administered at baseline, and then PRN based on retreatment criteria monthly from month 1 to 11.
  2. PDT:PRN PDT combination with conbercept injection based on retreatment criteria from month 3 to 11.
  PDT treatment must be administered within 7 days after the injection. If same day treatment of conbercept and PDT is performed, conbercept injection is to be administered at least 2 hours after the PDT.
  PDT should cover the whole area of polyps and branch vascular net (BVN).The PRN PDT retreatment intervals should be no less than 3 months.
  Interventions: Drug: conbercept; Procedure: Delayed PDT

INTERVENTIONS:
Drug: conbercept — At baseline conbercept injection is administered.And thereafter is administered based on re-treatment criteria from month 1 to 11.The PRN conbercept re-injection should be monthly.
  Other Names: lumitin
Procedure: Initial PDT — At baseline PDT with verteporfin is administered initially.And thereafter PDT is administered based on re-treatment criteria from month 3 to 11.The PRN PDT retreatment intervals should be no less than 3 months.
  Other Names: verteporfin
  Arms: Initial PDT combination with Conbercept
Procedure: Delayed PDT — PDT is administered based on re-treatment criteria from month 3 to 11.The PRN PDT retreatment intervals should be no less than 3 months.
  Other Names: verteporfin
  Arms: Delayed PDT combination with Conbercept

SUMMARY:
To compare the initial versus delayed verteporfin photodynamic therapy (PDT) in combination with conbercept in patients with symptomatic polypoidal choroidal vasculopathy (PCV).

DETAILED DESCRIPTION:
Polypoidal choroidal vasculopathy (PCV) is characterized by polypoidal choroidal vascular dilatation with or without abnormally branching vascular networks(BVN) on indocyanine green angiography (ICGA). It has been considered to be a subtype of wet age-related macular degeneration(wAMD). PCV is more prevalent in Asian patients than in white patients; nearly half of Chinese patients who was diagnosed with wAMD actually was PCV.

However, recently, the first choice treatment for wAMD has shifted to anti-vascular endothelial growth factor (VEGF) drugs, such as bevacizumab(Avastin,Genentech Inc), ranibizumab (Lucentis, Genentech Inc)and aflibercept (Eylea, Regeneron,Berlin,Germany) from PDT, and the vision improving effect has been confirmed regardless of race or disease subtype. Therefore, eyes with PCV can be treated initially with anti-VEGF drugs, however, they are limited in their ability to resolve polypoidal lesions, for which PDT works effectively.

Combination therapy of PDT and anti-VEGF drugs provides the complementary effects of both treatments, but it remains unknown whether PDT should have been administered at the beginning of treatment or during follow-up of anti-VEGF therapy. The purpose of this study was to compare the 12-months treatment results of initial and delayed PDT combined with conbercept (Lumitin, Chengdu Kang Hong Biotech Co., Ltd., Sichuan, China) for PCV.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender，age ≥ 40.
2. BCVA at study entry of 34 to 79 letters (Snellen Equivalent 20/200 to 20/25).
3. Naive symptomatic PCV patients.
4. Presence of PCV assessed based on ICG with active polyps with or without abnormal vascular network.
5. No refractive media opacity or small pupil narrow that influence the fundus examination.
6. Women must be using effective contraception, be post-menopausal for at least months prior to trial entry, or surgically sterile.
7. Ability to provide written informed consent and to return for all study visits.

Exclusion Criteria:

1. Active inflammation or infection in the study eye.
2. Uncontrolled intraocular pressure (>25 mmHg) in the study eye.
3. Ocular condition in the study eye which may impact vision and confound study outcomes (e.g. vitreomacular traction, epiretinal membrane with BCVA impact, ocular inflammation, retinal vascular diseases like diabetic retinopathy or diabetic macular edema).
4. Presence of centro macular scarring or atrophy indicating irreversible BCVA loss.
5. Prior treatment of the study eye with anti-VEGF therapy or systemic use of anti-VEGF products within 3 months prior to the study entry.
6. Previous vitrectomy, macular laser treatment, PDT, or intraocular steroids in the study eye.
7. Allergy to fluorescein, ICG, iodine, shellfish.
8. Pregnant or breast-feeding women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) in each group,Compare the difference between the two groups. | from baseline (month 0) to month 12

SECONDARY OUTCOMES:
The proportion of polyps regression assessed by ICGA in each group.Compare the difference between the two groups. | from Baseline (month 0) to month 12
Change in the Central Retinal Thickness (CRT), assessed by Spectral Domain-Optical Coherence Tomography (SD-OCT) | from Baseline baseline (month 0) to month 12
Total number of treatments with PDT and conbercept respectively | from Baseline (month 0) to month 12
Change in Best Corrected Visual Acuity (BCVA) at month 3 | from Baseline baseline (month 0) to month 3
Polyps regression, assessed by Indocyanine Green Angiography (ICGA) | from baseline (month 0) to month 3
Change in the Central Retinal Thickness (CRT), assessed by Spectral Domain-Optical Coherence Tomography (SD-OCT) | from baseline (month 0) to month 3
Frequency and severity of ocular and non-ocular adverse events over time. | from baseline (month 0) to month 12

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Liu, Professor, Principal Investigator — The Eye Hospital of Wenzhou Medical University
Locations (3):
- China (3):
  - The first affiliated hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yannuzzi LA, Sorenson JA, Guyer DR, Slakter JS, Chang B, Orlock D. Indocyanine green videoangiography: current status. Eur J Ophthalmol. 1994 Apr-Jun;4(2):69-81. doi: 10.1177/112067219400400201. PMID 7950339
- [Background] Yannuzzi LA, Ciardella A, Spaide RF, Rabb M, Freund KB, Orlock DA. The expanding clinical spectrum of idiopathic polypoidal choroidal vasculopathy. Arch Ophthalmol. 1997 Apr;115(4):478-85. doi: 10.1001/archopht.1997.01100150480005. PMID 9109756
- [Background] Yannuzzi LA, Wong DW, Sforzolini BS, Goldbaum M, Tang KC, Spaide RF, Freund KB, Slakter JS, Guyer DR, Sorenson JA, Fisher Y, Maberley D, Orlock DA. Polypoidal choroidal vasculopathy and neovascularized age-related macular degeneration. Arch Ophthalmol. 1999 Nov;117(11):1503-10. doi: 10.1001/archopht.117.11.1503. PMID 10565519
- [Background] Ciardella AP, Donsoff IM, Huang SJ, Costa DL, Yannuzzi LA. Polypoidal choroidal vasculopathy. Surv Ophthalmol. 2004 Jan-Feb;49(1):25-37. doi: 10.1016/j.survophthal.2003.10.007. PMID 14711438
- [Background] Imamura Y, Engelbert M, Iida T, Freund KB, Yannuzzi LA. Polypoidal choroidal vasculopathy: a review. Surv Ophthalmol. 2010 Nov-Dec;55(6):501-15. doi: 10.1016/j.survophthal.2010.03.004. Epub 2010 Sep 20. PMID 20850857
- [Background] Gomi F, Tano Y. Polypoidal choroidal vasculopathy and treatments. Curr Opin Ophthalmol. 2008 May;19(3):208-12. doi: 10.1097/ICU.0b013e3282fb7c33. PMID 18408495
- [Background] Laude A, Cackett PD, Vithana EN, Yeo IY, Wong D, Koh AH, Wong TY, Aung T. Polypoidal choroidal vasculopathy and neovascular age-related macular degeneration: same or different disease? Prog Retin Eye Res. 2010 Jan;29(1):19-29. doi: 10.1016/j.preteyeres.2009.10.001. Epub 2009 Oct 23. PMID 19854291
- [Background] Koh AH; Expert PCV Panel; Chen LJ, Chen SJ, Chen Y, Giridhar A, Iida T, Kim H, Yuk Yau Lai T, Lee WK, Li X, Han Lim T, Ruamviboonsuk P, Sharma T, Tang S, Yuzawa M. Polypoidal choroidal vasculopathy: evidence-based guidelines for clinical diagnosis and treatment. Retina. 2013 Apr;33(4):686-716. doi: 10.1097/IAE.0b013e3182852446. PMID 23455233
- [Background] Qu J, Cheng Y, Li X, Yu L, Ke X; AURORA Study Group. EFFICACY OF INTRAVITREAL INJECTION OF CONBERCEPT IN POLYPOIDAL CHOROIDAL VASCULOPATHY: Subgroup Analysis of the Aurora Study. Retina. 2016 May;36(5):926-37. doi: 10.1097/IAE.0000000000000875. PMID 26595362
- [Background] Gomi F, Oshima Y, Mori R, Kano M, Saito M, Yamashita A, Iwata E, Maruko R; Fujisan Study Group. INITIAL VERSUS DELAYED PHOTODYNAMIC THERAPY IN COMBINATION WITH RANIBIZUMAB FOR TREATMENT OF POLYPOIDAL CHOROIDAL VASCULOPATHY: The Fujisan Study. Retina. 2015 Aug;35(8):1569-76. doi: 10.1097/IAE.0000000000000526. PMID 25830698
- [Background] Koh A, Lee WK, Chen LJ, Chen SJ, Hashad Y, Kim H, Lai TY, Pilz S, Ruamviboonsuk P, Tokaji E, Weisberger A, Lim TH. EVEREST study: efficacy and safety of verteporfin photodynamic therapy in combination with ranibizumab or alone versus ranibizumab monotherapy in patients with symptomatic macular polypoidal choroidal vasculopathy. Retina. 2012 Sep;32(8):1453-64. doi: 10.1097/IAE.0b013e31824f91e8. PMID 22426346
- [Background] Oishi A, Kojima H, Mandai M, Honda S, Matsuoka T, Oh H, Kita M, Nagai T, Fujihara M, Bessho N, Uenishi M, Kurimoto Y, Negi A. Comparison of the effect of ranibizumab and verteporfin for polypoidal choroidal vasculopathy: 12-month LAPTOP study results. Am J Ophthalmol. 2013 Oct;156(4):644-51. doi: 10.1016/j.ajo.2013.05.024. Epub 2013 Jul 20. PMID 23876867
- [Derived] Sun Z, Gong Y, Yang Y, Huang Y, Yu S, Pei J, Lin B, Zhou R, Li Y, Li Y, Zhang J, Liu X. Efficacy of Initial vs. Delayed Photodynamic Therapy in Combination With Conbercept for Polypoidal Choroidal Vasculopathy. Front Med (Lausanne). 2022 Feb 9;8:791935. doi: 10.3389/fmed.2021.791935. eCollection 2021. PMID 35223882